CLINICAL TRIAL: NCT07144436
Title: Investigating the Feasibility, Efficacy, and Renormalization of Pain-Regulation Brain Circuits Underlying At-Home Transcutaneous Auricular Neuromodulation (tAN) for Managing Chronic Post-Stroke Pain
Brief Title: Post-stroke Pain tAN-fMRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Xiaolong Peng, Research Instructor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00145968
Record Dates: First submitted 2025-08-13; First posted 2025-08-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Post Stroke Pain
Keywords: Pain; Stroke
MeSH Terms: conditions — Pain; Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2 Weeks Sham tAN followed by 2 Weeks Active tAN (Experimental): Participants will be randomized to receive 2 weeks of at-home, self-administered sham Transcutaneous Auricular Neurostimulation (tAN), followed by 2 weeks of at-home, self-administered active Transcutaneous Auricular Neurostimulation (tAN).
  Interventions: Device: Transcutaneous Auricular Neurostimulation
- Four Weeks of Active Transcutaneous Auricular Neurostimulation (Experimental): Participants will be randomized to receive 2 weeks of at-home, self-administered active Transcutaneous Auricular Neurostimulation (tAN), followed by 2 additional weeks of at-home, self-administered active Transcutaneous Auricular Neurostimulation (tAN).
  Interventions: Device: Transcutaneous Auricular Neurostimulation

INTERVENTIONS:
Device: Transcutaneous Auricular Neurostimulation — Transcutaneous Auricular Neurostimulation (tAN) is a wearable, electrical stimulation device that delivers electricity to specific parts of the human ear.

SUMMARY:
The purpose of this study is to explore whether 4 weeks of at-home transcutaneous auricular neurostimulation (tAN) can reduce chronic pain after a stroke. Investigators will recruit up to 24 participants with chronic post-stroke upper extremity pain. The goal is to determine if there is a pain reduction after ear stimulation.

DETAILED DESCRIPTION:
In this study, the investigators main goal is to establish transcutaneous auricular neurostimulation (tAN) as an effective non-invasive neuromodulation method for pain management of post-stroke pain (PSP) and to investigate the brain circuit changes between pre- and post-treatment in individuals with PSP using brain imaging techniques.

Aim 1. Assess the feasibility and efficacy of self-administered, at-home tAN for pain management in stroke survivors with chronic pain compared to sham.

Aim 2. Investigate pain-induced brain activity changes over a one-month tAN treatment to understand the analgesic mechanisms of tAN.

Aim 3. Explore renormalization of brain functional connectivity and dynamic brain state throughout tAN treatment and develop brain imaging biomarkers to track and predict treatment efficacy for chronic post-stroke pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Have the capacity and ability to provide one's own consent in English and sign the informed consent document.
* Ischemic or hemorrhagic stroke that occurred at least 6 months prior

Exclusion Criteria:

* Primary intracerebral hematoma or subarachnoid hemorrhage
* Documented history of dementia
* Documented history of uncontrolled depression or psychiatric disorder
* Uncontrolled hypertension despite treatment, specifically SBP (Systolic Blood Pressure) / DBP (Diastolic Blood Pressure) >=180/100mmHg
* Contraindicated for MRI scanning
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensory Threshold | 4 weeks
  We will determine the pain threshold with a 30 × 30 mm thermode attached to the non-affected forearm of participants (TSA2 thermode; Medoc, Durham, NC, USA). Using the TSA2, we will determine heat sensitivity beginning at 32°C and increasing by 0.5°C per second. Participants will be asked to press a button (to record temperatures) when the stimulus is first detected (sensory threshold). We will acquire QST data at baseline, after one session (30 minutes) of tAN, after 2 weeks of tAN, and after 4 weeks of tAN.
Pain Threshold | 4 weeks
  We will determine the pain threshold with a 30 × 30 mm thermode attached to the non-affected forearm of participants (TSA2 thermode; Medoc, Durham, NC, USA). Using the TSA2, we will determine heat sensitivity beginning at 32°C and increasing by 0.5°C per second. Participants will be asked to press a button (to record temperatures) when the stimulus becomes painful (pain threshold). We will acquire QST data at baseline, after one session (30 minutes) of tAN, after 2 weeks of tAN, and after 4 weeks of tAN.
Pain tolerance | 4 weeks
  We will determine the pain threshold with a 30 × 30 mm thermode attached to the non-affected forearm of participants (TSA2 thermode; Medoc, Durham, NC, USA). Using the TSA2, we will determine heat sensitivity beginning at 32°C and increasing by 0.5°C per second. Participants will be asked to press a button (to record temperatures) when the stimulus is intolerable (pain tolerance). We will acquire QST data at baseline, after one session (30 minutes) of tAN, after 2 weeks of tAN, and after 4 weeks of tAN.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Peng, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - 30 Bee Street, Charleston, South Carolina
  - Medical University of South Carolia, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
De-identified imaging, behavioral, and QST data may be shared in aggregate or via secure repositories for future research.